CLINICAL TRIAL: NCT04533373
Title: The Effect of DIEP Flap Neurotization on Sensory Restoration After Breast Reconstruction
Brief Title: Sensory Restoration After DIEP Flap Neurotization
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB expired
Sponsor: Johns Hopkins University (Other)
Collaborators: Axogen Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00167074
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Breast Reconstruction; Sensory Restoration
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurotized Patients (Experimental): Neurotization will be performed at the time of reconstruction.
  Interventions: Procedure: DIEP Flap Neurotization
- Non-Neurotized Patients (No Intervention): No Neurotization will be performed at the time of reconstruction.

INTERVENTIONS:
Procedure: DIEP Flap Neurotization — We will be performing breast reconstruction using tissue from the patient's abdomen and transferring it to the chest wall to repair the mastectomy defect. Sensory function is restored by using the nerve that supplies the skin of this abdominal tissue (i.e the new "source") that is being transferred and attaching it to a nerve in the chest wall.
  Arms: Neurotized Patients

SUMMARY:
Common goals of breast reconstruction include obtaining satisfactory breast symmetry, softness, and appropriate size and shape. Advances in surgical techniques have prompted a new goal: achieving breast sensation after reconstructive surgery. This desire has led the surgical community to investigate operative techniques for achieving this goal. However, few studies have examined the effectiveness of breast sensory restoration.

Sensory nerves are nerves responsible for sensation from skin. When a sensory nerve is cut, sensation is lost to the area supplied by the nerve. In the case of Breast reconstruction this involves the nerves supplying the skin overlying breast(s). 'Neurotization' refers to regeneration of the nerve after it has been cut. This means that the cut nerve is being repaired in order to restore its function. In Neurotization this repair is carried out using a new "source". In this case, the investigators want to restore function of the nerves that supply the skin overlying the breast(s).

The investigators will be performing breast reconstruction using tissue from the patient's abdomen and transferring it to the chest wall to repair the mastectomy defect. Sensory function is restored by using the nerve that supplies the skin of this abdominal tissue (i.e the new "source") that is being transferred and attaching it to a nerve in the chest wall.

The Avance® Nerve graft is a nerve graft material that has been produced by Axogen, Inc. The graft is made by processing donated human nerves. This graft is used during neurotization to bridge the gap and join the nerve from the abdominal tissue to the nerve in the chest wall. The use of the graft helps the body to attach these 2 nerves and improves nerve repair.

When neurotization is done without the nerve graft there is a possibility that the surgeon may require extra nerve material to join the 2 nerves. Traditionally, in this case the surgeon would have to obtain a separate donor nerve from another part of the patient's body. This technique carries the risk of complications to part of the body that the separate donor nerve was obtained from - loss of sensation, infection or neuroma formation (an abnormal growth of nerve tissue that can cause pain, burning or tingling sensation, numbness). The Avance nerve graft avoids the need for the additional donor nerve and the possible complications associated with it.

The Avance® Nerve Graft is currently being used in some women during breast reconstruction surgery, however the effectiveness of this procedure in improving the restoration of sensation has not been proven.

Women undergoing reconstruction of one breast and at the same time using the women's own tissue as part of standard clinical care, may join.

ELIGIBILITY:
Inclusion Criteria:

1. All patients presenting to Johns Hopkins who have had or will have mastectomy (therapeutic or prophylactic) and are planning to undergo unilateral mastectomy followed by breast reconstruction with autologous deep inferior epigastric perforator flap (DIEP) will be included.

   These patients will then be randomized in either of two treatment modalities:
   * Treatment Modality 1: Breast reconstruction with DIEP flap and neurotization.
   * Treatment Modality 2: Breast reconstruction with DIEP flap but without neurotization.
2. 18 years of age and older
3. The patient is aware of the nature of her malignancy if a malignancy has been diagnosed; understands the study purpose, requirements, and risks; and is able and willing to sign an informed consent.

Exclusion Criteria:

1. Autologous reconstruction where the flap is buried.
2. Exclusion criteria will encompass any patient with: diabetic neuropathy, thyroid disorders, collagen vascular disease, alcoholism, pernicious anemia, or any other severe underlying peripheral neuropathy including chemotherapy-induced neuropathy or neuropathy induced by other medications.
3. Pregnant or lactating women will be excluded from this study.
4. Women with recurrent breast cancer will be excluded.
5. Women with previous reconstructive procedures or who have previously undergone lumpectomy with radiation will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
12-month Breast sensation as assessed by the AcroValTM device | 12-months after DIEP Flap neurotization
  Breast sensation, measured in cutaneous thresholds using the AcroValTM device.

SECONDARY OUTCOMES:
Breast sensation at 6 months as assessed by the AcroValTM device | 6 months after DIEP flap breast reconstruction
  Breast sensation, measured in cutaneous thresholds using the AcroValTM device.
Breast sensation at 18 months as assessed by the AcroValTM device | 18 months after DIEP flap breast reconstruction
  Breast sensation, measured in cutaneous thresholds using the AcroValTM device.
Breast sensation at 24 months as assessed by the AcroValTM device | 24 months after DIEP flap breast reconstruction
  Breast sensation, measured in cutaneous thresholds using the AcroValTM device.
Breast-specific health-related quality of life using the Breast-Q® | 6 months after DIEP flap breast reconstruction
  The Breast-Q® is a validated patient reported outcomes questionnaire used to assess Breast specific patient satisfaction and Health-related quality of life. The Breast-Q is comprised of 2 domains - i) Satisfaction domains and ii) Well-being domains, which are further divided into sub-domains. We will be using 3 satisfaction sub-domains:
  i) Satisfaction with breasts ii) Satisfaction with Nipple iii) Satisfaction with outcome
  and 3 well-being sub-domains:
  i) Psychosocial well-being ii) Sexual well-being and iii) Physical well-being
  Each sub-domain will be scored on a scale of 0-100, where higher scores will indicate higher satisfaction.
Breast-specific health-related quality of life using the Breast-Q® | 12 months after DIEP flap breast reconstruction
  The Breast-Q® is a validated patient reported outcomes questionnaire used to assess Breast specific patient satisfaction and Health-related quality of life. The Breast-Q is comprised of 2 domains - i) Satisfaction domains and ii) Well-being domains, which are further divided into sub-domains. We will be using 3 satisfaction sub-domains:
  i) Satisfaction with breasts ii) Satisfaction with Nipple iii) Satisfaction with outcome
  and 3 well-being sub-domains:
  i) Psychosocial well-being ii) Sexual well-being and iii) Physical well-being
  Each sub-domain will be scored on a scale of 0-100, where higher scores will indicate higher satisfaction.
Breast-specific health-related quality of life using the Breast-Q® | 18 months after DIEP flap breast reconstruction
  The Breast-Q® is a validated patient reported outcomes questionnaire used to assess Breast specific patient satisfaction and Health-related quality of life. The Breast-Q is comprised of 2 domains - i) Satisfaction domains and ii) Well-being domains, which are further divided into sub-domains. We will be using 3 satisfaction sub-domains:
  i) Satisfaction with breasts ii) Satisfaction with Nipple iii) Satisfaction with outcome
  and 3 well-being sub-domains:
  i) Psychosocial well-being ii) Sexual well-being and iii) Physical well-being
  Each sub-domain will be scored on a scale of 0-100, where higher scores will indicate higher satisfaction.
Breast-specific health-related quality of life using the Breast-Q® | 24 months after DIEP flap breast reconstruction
  The Breast-Q® is a validated patient reported outcomes questionnaire used to assess Breast specific patient satisfaction and Health-related quality of life. The Breast-Q is comprised of 2 domains - i) Satisfaction domains and ii) Well-being domains, which are further divided into sub-domains. We will be using 3 satisfaction sub-domains:
  i) Satisfaction with breasts ii) Satisfaction with Nipple iii) Satisfaction with outcome
  and 3 well-being sub-domains:
  i) Psychosocial well-being ii) Sexual well-being and iii) Physical well-being
  Each sub-domain will be scored on a scale of 0-100, where higher scores will indicate higher satisfaction.
General health-related quality of life using the SF-12 | 6 months after DIEP flap breast reconstruction
  The SF-12 is a multipurpose short form (SF) survey with 12 questions, all selected from the SF-36 Health Survey. It has 2 components - i) Physical Health Composite score and ii) Mental Health Composite score. Each composite score is marked on a scale of 0-100, where a higher score indicates higher quality of life.
General health-related quality of life using the SF-12 | 12 months after DIEP flap breast reconstruction
  The SF-12 is a multipurpose short form (SF) survey with 12 questions, all selected from the SF-36 Health Survey. It has 2 components - i) Physical Health Composite score and ii) Mental Health Composite score. Each composite score is marked on a scale of 0-100, where a higher score indicates higher quality of life.
General health-related quality of life using the SF-12 | 18 months after DIEP flap breast reconstruction
  The SF-12 is a multipurpose short form (SF) survey with 12 questions, all selected from the SF-36 Health Survey. It has 2 components - i) Physical Health Composite score and ii) Mental Health Composite score. Each composite score is marked on a scale of 0-100, where a higher score indicates higher quality of life.
General health-related quality of life using the SF-12 | 24 months after DIEP flap breast reconstruction
  The SF-12 is a multipurpose short form (SF) survey with 12 questions, all selected from the SF-36 Health Survey. It has 2 components - i) Physical Health Composite score and ii) Mental Health Composite score. Each composite score is marked on a scale of 0-100, where a higher score indicates higher quality of life.
Change in breast sensation as assessed by the AcroValTM device | Baseline, 6, 12, 18 and 24 months after DIEP flap breast reconstruction
  Change in breast sensation from baseline, measured in cutaneous thresholds using the AcroValTM device.
Change in breast-specific health-related quality of life using the Breast-Q® | Baseline, 6, 12, 18, and 24 months after DIEP flap breast reconstruction
  The Breast-Q® is a validated patient reported outcomes questionnaire used to assess Breast specific patient satisfaction and Health-related quality of life. The Breast-Q is comprised of 2 domains - i) Satisfaction domains and ii) Well-being domains, which are further divided into sub-domains. We will be using 3 satisfaction sub-domains:
  i) Satisfaction with breasts ii) Satisfaction with Nipple iii) Satisfaction with outcome
  and 3 well-being sub-domains:
  i) Psychosocial well-being ii) Sexual well-being and iii) Physical well-being
  Each sub-domain will be scored on a scale of 0-100, where higher scores will indicate higher satisfaction.
Change in general health-related quality of life using the SF-12 | Baseline, 6, 12, 18, and 24 months after DIEP flap breast reconstruction
  The SF-12 is a multipurpose short form (SF) survey with 12 questions, all selected from the SF-36 Health Survey. It has 2 components - i) Physical Health Composite score and ii) Mental Health Composite score. Each composite score is marked on a scale of 0-100, where a higher score indicates higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Gedge D Rosson, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No